CLINICAL TRIAL: NCT01310868
Title: An Evaluation of the Tolerability and Feasibility of Combining 5-Amino-Levulinic Acid (5-ALA) With Carmustine Wafers (Gliadel) in the Surgical Management of Primary Glioblastoma (GALA-5 Trial)
Brief Title: Gliadel Wafer and Fluorescence-Guided Surgery With 5-ALA Followed by Radiation Therapy And Temozolomide in Treating Patients With Primary Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000696316; CRUK-UCL-09-0398 (Other Grant/Funding Number: Cancer Research UK and Samantha Dixon Brain Tumour Trust); 2010-022496-66 (EudraCT Number); 09/0398 (Other: University College London); 10/H0304/100 (Other: NRES Committee East of England - Cambridge East)
Record Dates: First submitted 2011-03-05; First posted 2011-03-09 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Aminolevulinic Acid; Carmustine; Radiotherapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-ALA and Gliadel wafers (Experimental): This is a single arm feasibility study to evaluate the safety and tolerability of combining 2 technologies (5-ALA and Gliadel wafers) in the surgical management of patients with GBM.
  Interventions: Drug: 5-ALA; Drug: Gliadel wafers; Radiation: Radiotherapy as normal based on standard clinical protocols determined by the neuro-oncologist; Drug: Concomitant chemotherapy as normal based on standard clinical protocols determined by the neuro-oncologist; Drug: Adjuvant chemotherapy as normal based on standard clinical protocols determined by the neuro-oncologist

INTERVENTIONS:
Drug: 5-ALA — 5-ALA is used to generate tumour specific fluorescence as an aid to surgical resection of GBM, prior to the insertion of Gliadel wafers
  Other Names: Amino-levulinic Acid; Gliolan
Drug: Gliadel wafers — The implantation of Carmustine Wafers (Gliadel) delivers carmustine- (3-bis 2-chloroethyl 1-1-nitrosourea (BCNU)) directly into the surgical cavity created after tumour resection.
  Other Names: Carmustine wafers; polifeprosan 20 with carmustine implant
Radiation: Radiotherapy as normal based on standard clinical protocols determined by the neuro-oncologist — 60Gy in 30 fractions (2Gy per fraction given once daily, five days per week (Monday-Friday) over 6 weeks. Radiotherapy delivered to gross tumour volume with 2-3cm margin. Standard treatment following neurosurgery for glioblastoma
Drug: Concomitant chemotherapy as normal based on standard clinical protocols determined by the neuro-oncologist — temozolomide given alongside the radiotherapy at 75mg/m2 daily from the first day of radiotherapy, until the last day of radiotherapy, but for no longer than 49 days. Standard treatment following neurosurgery for glioblastoma
Drug: Adjuvant chemotherapy as normal based on standard clinical protocols determined by the neuro-oncologist — Following a 4 week break after contomitant chemo/RT, temozolomide given 150-200mg/m2 TMZ 5/28 days for 6 cycles (dosage increase to 200mg/m2 on second and subsequent cycles dependent on haematological toxicity. Sites should follow local guidelines if different.). TMZ to be given on 5 consecutive days followed by 23 days with no TMZ, per cycle. Standard treatment following neurosurgery and concomitant chemo/RT for glioblastoma

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as Gliadel wafer and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy and temozolomide after surgery and Gliadel wafer may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects of fluorescence-guided surgery with 5-ALA given together with Gliadel wafer, followed by radiation therapy and temozolomide, in treating patients with primary glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish that the combined use of 5-ALA and Gliadel wafers during fluorescence-guided radical brain tumor resection is safe and does not compromise patients with primary glioblastoma from receiving or completing adjuvant standard radiotherapy plus temozolomide.

Secondary

* To gather preliminary evidence that the combined use of 5-ALA and Gliadel wafers at surgery has the potential to improve clinical outcome, via measurement of time to clinical progression.
* To gather preliminary evidence that this regimen at surgery has the potential to improve clinical outcome via measurement of survival at 24 months.

OUTLINE: This is a multicenter study.

Gliadel wafers are applied to resection cavity immediately after 5-ALA fluorescence-guided radical brain tumor resection. After recovery from surgery (within 6 weeks of surgery when possible ), patients receive adjuvant chemoradiotherapy comprising standard radiotherapy and temozolomide.

Tumor biopsy and blood sample may be collected at time of surgery for retrospective MGMT status analysis.

After surgery, patients are followed up at post-surgical visits, during subsequent therapy at routine clinic visits, and at 12, 18, and 24 months.

Peer reviewed and funded by Cancer Research UK.

ELIGIBILITY:
INCLUSION CRITERIA

i. The patient is reviewed at a specialist neuro-oncology multi-disciplinary team (MDT).

ii. Stealth MRI (neuronavigation) will be performed prior to surgery.

iii. Imaging is evaluated by a neuro-radiologist and judged to have typical appearances of a primary GBM

iv. Radical resection is judged to be realistic by the neurosurgeons at the MDT (i.e. NICE criteria for the use of Carmustine wafers can be met)

v. WHO performance status 0 or 1

vi. Age ≥18

vii. Patient judged by MDT to be fit for standard radical aggressive therapy for GBM (resection followed by RT with concomitant and adjuvant temozolomide)

EXCLUSION CRITERIA

i. GBM thought to be transformed low grade or secondary disease

ii. The patient has not been seen by a specialist MDT.

iii. There is uncertainty about the radiological diagnosis

iv. 5-ALA or Carmustine wafers is contra-indicated (inc known or suspected allergies to 5-ALA or porphyrins, or acute or chronic types of porphyria)

v. Pregnant or lactating women

vi. Known or suspected HIV or other significant infection or comorbidity that would preclude radical aggressive therapy for GBM

vii. Active liver disease (ALT or AST ≥5 x ULRR)

viii. Concomitant anti-cancer therapy except steroids

ix. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years

x. Previous brain surgery (including biopsy) or cranial radiotherapy

xi. Platelets <100 x109/L

xii. Mini mental status score <15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Watts, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (10):
- United Kingdom (10):
  - Addenbrooke's Hospital, Cambridge, England
  - Royal Preston Hospital, Preston, Lancashire
  - Ninewells Hospital, Dundee
  - Southern General Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - The Walton Centre, Liverpool
  - King's College Hospital, London
  - University College London Hospital/ National Hospital for Neurology and Neurosurgery, London
  - Royal Hallamshire Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study entry was based on imaging that has been judged to have typical appearances of a primary glioblastoma multiforme (GBM). Patients would have neurosurgery and GBM would be confirmed peri/post-operatively. If not GBM patients OR wafers+ 5-ala not administered then remain in the trial for follow up but were not included in the final analysis.
Period: Overall Study
Arm/Group | 5-ALA and Gliadel Wafers
Started | 72
Completed | 59
Not Completed | 13
Not completed — Do not have histologically confirmed GBM | 13

BASELINE CHARACTERISTICS:
Arm/Group | 5-ALA and Gliadel Wafers
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 49
Region of Enrollment [Number; unit: participants]
  United Kingdom | 72

OUTCOME MEASURES:

1. Primary Outcome: Safety, Tolerability, and Feasibility of Combination Intra-operative 5-ALA and Gliadel Wafers Prior to Adjuvant Radiotherapy Plus Temozolomide
Description: Procedure compliance: Proportion of 5-ALA resected patients who received Carmustine wafer implants (e.g to take into account rates of patients who did not receive Carmustine wafer implants due to 1) ventricular breach, 2) inaccurate peri-operative diagnosis, 3) intra-operative surgical decision)
  * Post-operative complication rate: Proportion of patients with a new post-operative deficit or surgical complication (wound infection, CSF leakage, intracranial hypertension)
  * No. of patients with chemoRT delay (i.e number who do not begin chemoRT 6 weeks after surgery) due to surgical complications*
  * No. of patients failing to start chemoRT due to surgical complications rather than tumour progression
  * No. of patients failing to complete chemoRT without interruption (RT with concomitant chemotherapy, and RT with concomitant plus adjuvant chemotherapy)
  * Proportion of patients with a lower WHO performance status after surgery with Carmustine wafers (at first post-operative clinic visit)
Time Frame: Date of surgery to end of temozolomide and radiotherapy treatment (up to 34 weeks)
Population: of 72 patients recruited, 62 received 5-ALA and carmustine wafers. Of these 62 patients, 59 were found to be eligible and included in the final analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 5-ALA and Gliadel Wafers
Number analyzed (Participants) | 72
Participants
  5-ALA resected patients receiving carmustine wafer | 62
  No. patients with post-op complications: number analyzed (Participants) | 59
  No. patients with post-op complications | 9
  No. Patients with chemoRT delay: number analyzed (Participants) | 59
  No. Patients with chemoRT delay | 6
  No. pts failing to complete uninterrupted chemoRT: number analyzed (Participants) | 59
  No. pts failing to complete uninterrupted chemoRT | 45
  no. pts w decr perform status after 5ala/carmustin: number analyzed (Participants) | 59
  no. pts w decr perform status after 5ala/carmustin | 27
  no. pts not starting chemoRT due to surgical comp: number analyzed (Participants) | 59
  no. pts not starting chemoRT due to surgical comp | 2

2. Secondary Outcome: Time to Clinical Progression
Time Frame: from the date of surgery to the date of the first MRI scan fitting the criteria for progression, or the date the clinical detrioration or death was first reported
Population: Patients receiving 5-ala and carmustine wafers during surgical resection for glioblastoma multiforme that was confirmed peri/post-operatively
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5-ALA and Gliadel Wafers
Number analyzed (Participants) | 59
months | 9.5 [7.5 to 9.8]

3. Secondary Outcome: Survival at 24 Months
Time Frame: from the date of surgery to 24 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5-ALA and Gliadel Wafers
Number analyzed (Participants) | 59
months | 15 [11.9 to 17.3]

ADVERSE EVENTS:
Arm/Group | 5-ALA and Gliadel Wafers
Serious Adverse Events (participants affected / at risk) | 26/59
Other Adverse Events (participants affected / at risk) | 23/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-ALA and Gliadel Wafers (N=59)
Wound dehiscence (Injury, poisoning and procedural complications) | 1
hematoma (Vascular disorders) | 1
thromboembolic event (Vascular disorders) | 3
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
cerebral spinal fluid leak (Nervous system disorders) | 2
headache (Nervous system disorders) | 1
stroke (Nervous system disorders) | 1
vasovagal reaction (Nervous system disorders) | 1
retinal detachment (Eye disorders) | 1
fever (General disorders) | 1
psychiatric disorders - other (steroid induced aggression) (Psychiatric disorders) | 1
colonic perforation (Gastrointestinal disorders) | 1
other - bowel perforation (Gastrointestinal disorders) | 1
intra-abdomial hemorrhage (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
muscle weakness left sided (Musculoskeletal and connective tissue disorders) | 1
infection - cerebral abscess (Infections and infestations) | 1
infections other (not specified) (Infections and infestations) | 2
sepsis (Infections and infestations) | 2
urinary tract infection (Infections and infestations) | 1
wound infection (Infections and infestations) | 2
seizure (Nervous system disorders) | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-ALA and Gliadel Wafers (N=59)
wound infection (Injury, poisoning and procedural complications) | 3
thrombolytic event (Vascular disorders) | 4
neutrophil count decreased (Investigations) | 4
platelet count decreased (Investigations) | 4
white blood cell decreased (Investigations) | 3
seizure (Nervous system disorders) | 5
lethargy (Nervous system disorders) | 3
nausea (Gastrointestinal disorders) | 4
vomiting (Gastrointestinal disorders) | 3
muscle weakness (Musculoskeletal and connective tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.